CLINICAL TRIAL: NCT06665191
Title: Prevalence of Tooth Wear, Predictive Risk Factors and Its Association with Oral Health-related Quality of Life Among Middle -aged Adult Patients Attending Dental Educational Hospital At Cairo University: Cross-sectional Study
Brief Title: Prevalence of Tooth Wear and Its Association with Oral Health-related Quality of Life
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Abdel-Latif Amin, Assistant lecturer, Cairo University
Other Study IDs: 1441991
Record Dates: First submitted 2024-10-09; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Tooth Wear; Attrition; Erosion
Keywords: Tooth wear; attrition; BEWE; Basic erosive wear examination; quality of life
MeSH Terms: conditions — Tooth Wear | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Middle aged Adults NOT suffering from dental wear: Middle aged Adults NOT suffering from dental wear attending dental educational hospital in Cairo University
- Middle aged adults Suffering from dental wear: Middle aged adults Suffering from dental wear attending dental educational hospital in Cairo University
  Interventions: Other: No Intervention: Observational study for prevalence of dental wear and its association with quality of life

INTERVENTIONS:
Other: No Intervention: Observational study for prevalence of dental wear and its association with quality of life — not applicable as it is an observational study testing the prevalence of dental wear in patients attending Cairo University
  Groups: Middle aged adults Suffering from dental wear

SUMMARY:
The aim of this study is to detect the prevalence of tooth wear (All forms of cumulative surface loss of mineralized tooth substance loss due to physical and chemico-mechanical process according to the definition of the European Organization for Caries Research (ORCA) and the International Cariology Research Group for Dental Research (IADR) i.e.: attrition, erosion and abrasion) among middle aged adult patients attending educational hospital at the Faculty of Dentistry, Cairo University and to analyze the distribution of lesions by gender and age, frequency of acidic foods and drinks consumption, medicine usage, chewing habits, systemic diseases, tooth brushing habits, and family socio economic status. Moreover, to evaluate the quality of life among middle aged elderly patients in relation to existence of tooth wear.

The study focuses on middle-aged adult patients (31-45 years) attending the Faculty of Dentistry at Cairo University during 2025-2026. It is an analytical cross-sectional study aimed at assessing the prevalence and risk level of tooth wear using the Basic Erosive Wear Examination Index (BEWE). The BEWE categorizes tooth wear into four levels (0 = no wear, 3 = severe wear), and risk levels are determined by the cumulative score.

Primary outcome: the prevalence of tooth wear and associated risk levels. Secondary outcomes: identifying predictive risk factors and assessing the Oral Health Impact Profile (OHIP) for patients diagnosed with tooth wear. All participants will be examined, and those with a BEWE score above 0 will be considered affected. Risk levels will be stratified as no risk, low, medium, or high.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients whose age between 31 to 45 years old. 2- Egyptian 3- Males & Females 4- Provide informed consent 5- Ability to comprehend asked questions

Exclusion Criteria:

* 1- Patients under or over the selected age group 2- Patients using fixed orthodontic appliances, 3- Patients with special needs

Ages: 31 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Middle aged adult patient attending educational hospital for dental treatments free of charfge
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Prevalence and risk level of tooth wear | 1 year
  Prevalence of wear will be tested using Basic erosive wear examination index (BEWE) 0 =no tooth wear
  1. =minimal loss of surface texture
  2. = distinct defect, hard tissue loss <50% of the surface area
  3. = hard tissue loss ≥ 50% of the surface area The examination is repeated for all teeth in a sextant but only the surface with the highest score is recorded for each sextant.
  To calculate prevalence Examined participants with score 0 will represent unaffected population % Examined participants with scores above 0 will represent the affected population % Stratification of risk levels will be done for affected population according to BEWE risk levels. The sum of the scores is calculated to provide the BEWE risk level (0-14) 0-2 = no risk 3-8= low risk 9-13= medium risk 14= high risk

SECONDARY OUTCOMES:
• Predictive risk factors for all participants using a questionnaire | 1year
  Sociodemographic data:
  age, gender, occupation and education
  Predictive risk factors:
  1. Frequency of consuming acidic food and fruits, carbonated beverages and alcohol.
  2. Medicine usage ( vitamin c, aspirin)
  3. Chewing habits
  4. Systemic diseases
  5. Tooth brushing habits
  6. Family socio economic status.
Oral Health-Related Quality of Life (OHRQoL) using a questionnaire | 1 year
  OHRQoL will be measured using Oral Health Index Profile (OHIP-14) questionnaire
  OHIP-14 is a 14-item questionnaire that measures :
  Functional limitation Physical pain Phycological discomfort Physical disability Social disability Phycological disability Handicap
  It measures responses on a Likert scale (0-4) with the following values:
  Never (0) Hardly ever (1) Occasionally (2) Frequently (3) Very frequently (4) Points for each response are summed so that each patient can score a minimum of 0 points and a maximum of 56 points. Low scores indicate better self-perceived quality of life, and high scores indicate worse self-perception of oral quality of life Participants diagnosed with tooth wear

IPD SHARING:
Plan to Share IPD: Undecided